CLINICAL TRIAL: NCT00523354
Title: Phase 2 Proof-of-Concept Study to Analyze the Efficacy of in TNF-Alpha Blockade in Adult Patients With Severe, Corticosteroid-Dependent Eosinophilic Esophagitis
Brief Title: Off Label Use of Infliximab in Adult Patients With Severe Eosinophilic Esophagitis
Acronym: IEE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss EE Study Group (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Swiss EE-Study Group
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Esophagitis
Keywords: Eosinophilic Esophagitis; TNF-alpha; TNF-alpha Blockade; Infliximab
MeSH Terms: conditions — Esophagitis; Eosinophilic Esophagitis | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (open-label) (Experimental): prospective, open label, uncontrolled trial
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Induction therapy with 2 infusions, each 5 mg/kg body weight within 2 wks
  Other Names: Remicade

SUMMARY:
Eosinophilic Esophagitis (EE) is a chronic inflammatory disorder of the esophagus with a constantly increasing prevalence. It has been demonstrated that the expression of the cytokine TNF-α is up regulated in EE and that this pro-inflammatory cytokine is highly expressed by the keratinocytes of the esophageal epithelium in patients with active EE. Furthermore, it has been shown that TNF-α is capable to induce eotaxin-3 production in keratinocytes. These results suggest that TNF-α plays a crucial role in the pathogenesis of EE. Based on these findings, the investigators plan a prospective T1 translational study with the purpose to evaluate the efficacy of an Infliximab monotherapy in adult patients with severe, corticosteroid-dependent EE.

DETAILED DESCRIPTION:
Study Principle: An open-conducted, un-controlled, off label use of Infliximab will be performed in at least 3 individuals with Eosinophilic Esophagitis (EE) to evaluate the efficacy of an TNF-α blockade in the treatment of adult patients with severe, isolated EE.

Rationale for this Trial: Eosinophilic Esophagitis is a chronic, TH2-type dominant inflammatory disorder of the esophagus with a constantly increasing prevalence. It has been demonstrated that the cytokines TNF-α and IL-5 as well as the chemokine eotaxin-3 play a crucial role in the immuno-pathogenesis of this disease. These mediators are potential targets for therapeutic interventions. The established diagnostic criteria of EE are PPI-resistent esophageal related symptoms in combination with an infiltration of the esophageal mucosa with more than 20 eosinophils/hpf, a tissue where eosinophils are not normally encountered.

Treatment strategies in chronic inflammations have basically two goals: 1) Relief of symptoms; and 2) Prevention of long-term damage of the affected organ, due to a persistence of an uncontrolled inflammation. Standard recommendations for medical therapy of EE include systemic or topical corticosteroids and leukotriene antagonists. The treatment with corticosteroids is limited by the occurence of steroid-dependence and steroid-resistance, as well as the corticosteroid adherent side effects.

Infliximab, a chimeric monoclonal IgG antibody, is a potent inhibitor of the soluble and the membrane-bound form of TNF-α. Its efficacy in inducing and maintaining a remission in several TH1- and TH2-type inflammations is well documented. Infliximab is since more than 5 years approved for the therapy of these immune-mediated inflammations. Today, it is used as standard therapy in a subset of severe forms in these disorders. Meanwhile an overwhelming mass of data has confirmed the efficacy and the safety of this compound.

Purpose of this Study:The purpose of this pilot-trial is to evaluate the efficacy of a TNF-α blockade with Infliximab monotherapy as induction-treatment in adult patients with severe EE.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with severe, corticosteroid-dependent eosinophilic esophagitis

Exclusion Criteria:

* Pregnancy
* Evidence of latent or active tuberculosis
* Other contra-indications for TNF-alpha blockers
* Unstable medical conditions
* Malignancies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-08; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Tissue eosinophilia before and after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Uwe Simon, MD and PhD, Study Chair — Deaprtment of Pharmacology, University Bern, Bern, Switzerland
Locations (1):
- EE-Clinics, Praxis Roemerhof, Olten, Canton of Solothurn, Switzerland